CLINICAL TRIAL: NCT01783002
Title: Pre-operative Parathyroid Imaging: a Comparison of 11C-Methionine PET, 18F-FDG PET AND SPEC-CT for the Detection of Hyperfunctional Parathyroid Tissues
Brief Title: 11C Methionine PET for the Detection of Hyperfunctional Parathyroid Tissues
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H12-01220
Record Dates: First submitted 2013-01-04; First posted 2013-02-04 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — carbon-11 methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary hyperparathyroidism (Experimental): Subjects with biochemical evidence, including elevated serum calcium and PTH levels, of primary hyperparathyroidism. All patients will undergo 11C-methionine PET/CT, SPECT-CT and 18F-FDG PET/CT scanning.
  Interventions: Radiation: 11C-Methionine PET/CT scanning; Radiation: 18F-FDG PET/CT scanning; Radiation: SPECT-CT scanning

INTERVENTIONS:
Radiation: 11C-Methionine PET/CT scanning — PET with the radiopharmaceutical carbon-11 methionine (11C-MET) has been considered to improve diagnosis due to a superior spatial resolution and higher specificity compared to other radiotracers such as 18F-FDG. For the 11C-MET PET/CT, the patient will receive an intravenous bolus injection of 11C-MET as manufactured at the BCCA production facility at a dose of 6 (0.16 mCi) MBq per kilogram but not to exceed 555 MBq (15 mCi).
  Other Names: 11C-MET
Radiation: 18F-FDG PET/CT scanning — For PET/CT scans, the patient will first receive an intravenous bolus injection of 18F-FDG as manufactured at the BCCA production facility in a dose determined by body weight but not to exceed 521 MBq (14.1 mCi). Our standard adult prescription (70kg adult) for 18F-FDG is 296 MBq (8.0 mCi). The target dose for body scans is increased by 59.2 MBq (1.6 mCi) for every 20 kg increase in body weight to a maximum target dose of 474 MBq (12.8 mCi).
Radiation: SPECT-CT scanning — For the SPECT-CT scan, each injection of intravenous 99mTc-MIBI is dosed at a maximum of 20 mCi (740MBq), as per usual standard of care. The energy window of each scan is at 140 keV, consistent with the standard of SPEC-CT imaging techniques.

SUMMARY:
The overall sensitivity and specificity of 11C-MET PET/CT is superior to 18F-FDG PET/CT and conventional SPECT-CT for the detection of abnormal parathyroid glands.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Primary: To compare the accuracy, sensitivity and specificity of 11C-methionine (MET) PET/CT and 99mTc-MIBI SPECT-CT in the detection of pathologic parathyroid glands in patients with primary hyperparathyroidism.

Secondary:To compare the accuracy, sensitivity and specificity of 11C-MET and 18F-FDG PET/CT scans in the detection of pathologic parathyroid glands in patients with primary hyperparathyroidism.

STUDY DESIGN A phase II diagnostic imaging, single-centre study to compare the accuracy of 11C-MET PET/CT with standard 99mTc-MIBI SPECT-CT and with 18F-FDG PET/CT imaging in patients with primary hyperparathyroidism.

STUDY POPULATION Number of Subjects: 50 patients Number of groups: 1: 50 with primary hyperparathyroidism. Age/Gender: Age greater than or equal to 19 years / Male and Female Study specific requirements: Subjects with clinically suspected primary hyperparathyroidism who require 99mTc-MIBI SPECT-CT parathyroid imaging.

INVESTIGATIONAL PRODUCT Product: 11C-Methionine Route of administration: Intravenous Dosage(s) and frequency: Radioactive dose of 11C-Methionine of 6 MBq per kilogram body weight per injection (maximum dose of 555 MBq); one injection per patient.

COMPARATOR PRODUCTS Product: 99mTc-Methoxyisobutylisonitrite; 18F-Fluorodeoxyglucose Route of administration: Intravenous Dosage(s) and frequency: (1) Radioactive dose of 99mTc-Methoxyisobutylisonitrite of 555 - 740 MBq per injection; one injection per patient. (2) Radioactive dose of 18F-Fluorodeoxyglucose of 296 - 521 MBq per injection; one injection per patient.

EVALUATION CRITERIA Efficacy: The comparison of the accuracy, sensitivity, and specificity of 11C-MET PET/CT with 99mTc-MIBI SPECT-CT and 18F-FDG PET/CT in the detection of pathologic parathyroid glands in patients with primary hyperparathyroidism.

Safety: Vital signs before and following 11C-MET administration; adverse events collection.

ELIGIBILITY:
Inclusion Criteria:

* Adults > age 18;
* Able to provide written informed consent;
* Subjects with biochemical evidence, including elevated serum calcium and PTH levels, of primary hyperparathyroidism.

Exclusion Criteria:

* Subjects with previous successful parathyroidectomy and parathyroid tissue reimplantation;
* Pregnancy;
* Subjects who are unable to tolerate the physical/logistical requirements of completing two PET/CT scans, including lying still for a prolonged period of time and receiving two intravenous injections.
* Subjects who exceed the safe weight limit of the PET/CT bed (204.5 kg) or who cannot fit through the PET/CT machine (diameter 70cm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
To compare the sensitivity of 11C-MET PET/CT, SPECT-CT and 18F-FDG PET/CT in the detection of pathologic parathyroid glands in patients with primary hyperparathyroidism | Patient will undergo the scans at baseline
  Sensitivity is the percentage of patients that were correctly identified to have an abnormal parathyroid gland by the imaging studies.
To compare the specificity of11C-MET PET/CT, SPECT-CT and 18F-FDG PET/CT in the detection of pathologic parathyroid glands in patients with primary hyperparathyroidism | Patient will undergo the scans at baseline
  Specificity is defined as the percentage of patients that were correctly rejected for having an abnormal parathyroid gland by the imaging studies.

SECONDARY OUTCOMES:
To evaluate the safety profile of 11C-MET PET/CT. | Up to 2 weeks
  All adverse events will be recorded. An Adverse Event (AE) is any untoward, undesired, unplanned medical occurrence in a participant and does not necessarily have a causal relationship with the study intervention. Expected adverse events from PET/CT scans include bruising, bleeding or infection at the site of intravenous radiotracer injection. Other expected adverse events include feeling of discomfort or claustrophobia from being in the scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Anderson, MD, FRCSC, Principal Investigator — University of British Columbia; Vancouver General Hospital; Don Wilson, MD, FRCPC, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada